CLINICAL TRIAL: NCT04925973
Title: Tofacitinib for Hospitalized Acute Severe Ulcerative Colitis Management (the TRIUMPH Study)
Brief Title: Tofacitinib for Hospitalized Acute Severe Ulcerative Colitis Management
Acronym: TRIUMPH
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: University of Manitoba (Other); University of British Columbia (Other); McGill University (Other); University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11428
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Ulcerative Colitis Acute
MeSH Terms: interventions — tofacitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment arm (Experimental): Tofacitinib 10mg PO BID
  Interventions: Drug: Tofacitinib 10 MG [Xeljanz]

INTERVENTIONS:
Drug: Tofacitinib 10 MG [Xeljanz] — Tofacitinib 10mg PO BID

SUMMARY:
The TRIUMPH study was designed to build on the existing literature by studying the efficacy of tofacitinib in hospitalized patients with acute severe ulcerative colitis. This trial will provide evidence for a possible new indication for the use of tofacitinib.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18 to 75 with ulcerative colitis (either known UC based on prior history with histological confirmation or new diagnosis)
2. Symptoms consistent with severe acute ulcerative colitis as defined by modified Truelove and Witts score (MTWSI) > 10 points
3. Primary non-response or secondary loss of response to anti-TNFα/anti-integrin therapies/anti-interleukin therapies OR immunomodulators OR non-response to minimum 3 days and maximum of 7 days of intravenous corticosteroids (intravenous at dose equivalent of prednisone 50mg daily / methylprednisolone 40mg daily).

   a. For patients using anti-TNFα or anti-integrin or anti-interleukin therapies, they must have been on a stable dose of one of the following: i. Adalimumab in the 14 days prior to screening ii. Golimumab in the 28 days prior to screening iii. Infliximab in the 28 days prior to screening iv. Vedolizumab in the 28 days prior to screening v. Ustekinumab in the 28 days prior to screening b. Persons on biologic therapy will have drug levels drawn during the time of hospitalization
4. Able to provide written informed consent
5. Treatment with concomitant corticosteroids or 5-ASA products is permitted, however patients will be placed on a corticosteroid weaning regimen after initiating study protocols. For patients using biologics or immunomodulators, these will be discontinued prior to initiation of tofacitinib.

Exclusion Criteria:

1. Enteric infection confirmed before inclusion into study by stool microscopy, culture, or histology (including Clostridum difficile, Campylobacter, Salmonella, Shigella, Cytomegalovirus, Human Immunodeficiency Virus, Epstein Bar Virus)
2. Clinical signs of sepsis
3. Patient has indication for surgery instead of medical rescue therapy (ex. toxic megacolon, massive exsanguination, or perforation)
4. Positive blood (beta-HCG) pregnancy test or currently lactating, or women of childbearing potential not willing to use double barrier contraception for the duration of the active part of the study and for 4 weeks after the last dose of tofacitinib

   a. Participants will be sufficiently educated to ensure compliance with double barrier contraception prior to enrollment in the study
5. Current malignancy
6. Serious co-morbidity including but not limited to:

   a. Immunodeficiency b. Recent myocardial infarction or stroke (in the past month) c. History of heart, respiratory, renal, or hepatic failure i. Heart failure as defined as ejection fraction of <50% as determined by transthoracic echo ii. Respiratory failure as defined as PaO2 <60mmHg iii. Hepatic failure as defined as INR > 2.5 with total bilirubin >30 iv. Renal failure as defined as a creatinine clearance of 40ml/min (as estimated by the Cockroft-Gault equation) d. Infections such as abscess, opportunistic infection, or sepsis
7. English not adequate in absence of local translation service
8. Currently taking part in another clinical trial
9. Treatment with tofacitinib in the 3 months prior to screening
10. Use of strong CYP (3A4 or 2C19) inhibitors or inducers such as antifungals (ketoconazole, fluconazole), St John's wort or rifampin a. Patients will be told to avoid consumption of grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Clinical response at day 7 | 7 days
  To determine the effectiveness (combined and endoscopic response) and safety of tofacitinib in patients with acute severe UC who experience treatment failure to steroids or anti-TNFα/anti-integrin therapies/anti-interleukin therapies. The primary outcome of this study is to assess clinical response at day 7 among patients who receive tofacitinib. This will be determined by the percentage of patients who achieve clinical response at day 7 (MTWSI reduction 3 or more points and MTWSI < 10).

SECONDARY OUTCOMES:
1. Percentage of patients who achieve clinical remission at day 7, and weeks 12, 26, and 52 (Partial Mayo score < 2, with no subscore >1) | 52 weeks
Number of colectomies (emergency and planned) during the 52 weeks | 52 weeks
Number of patients requiring switch in therapy (i.e. initiation of another biological medication, start of a different clinical trial with another active drug, etc) during the 52 weeks | 52 weeks
Percentage of patients who achieve clinical response at weeks 12, 26, and 52 (MTWSI reduction 3 or more points and MTWSI < 10) | 52 weeks
For patients who have response, to determine the mean number of days before detection of clinically significant response (MTWSI reduction of 3 or more points) population. | 7 days
To determine the rate of corticosteroid-free clinical remission based on Number of patients with initial Mayo 2/3 disease at flexible sigmoidoscopy that achieve endoscopic improvement (Mayo score 0 or 1) at week 26 | Week 26
Comparison of absolute change from baseline endoscopic Mayo score at week 26 | Week 26
Comparison of number of patients with severe colitis based on histology who are able to achieve histological improvement (mild or inactive colitis) at week 26 | Week 26
Proportion of individuals who experience a severe adverse event over the course of treatment | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Narula, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will be collected from study sites and analyzed.

REFERENCES:
- [Derived] Narula N, Pray C, Hamam H, Peerani F, Hansen T, Bessissow T, Bressler B, Arun A, Schmit M, Castelli J, Marshall JK. Tofacitinib for Hospitalized Acute Severe Ulcerative Colitis Management (The TRIUMPH Study). Crohns Colitis 360. 2025 Feb 15;7(1):otaf013. doi: 10.1093/crocol/otaf013. eCollection 2025 Jan. PMID 40092634